CLINICAL TRIAL: NCT01201707
Title: The Effectiveness of Endovascular Treatment of Chronic Cerebrospinal Venous Insufficiency (CCSVI) in Patients With Multiple Sclerosis
Brief Title: Evaluation of Angioplasty in the Treatment of Chronic Cerebrospinal Venous Insufficiency (CCSVI) in Multiple Sclerosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inability to enroll adequate number of patients
Sponsor: Community Care Physicians, P.C. (Other)
Responsible Party: Principal Investigator, Gary Siskin, MD, Professor and Chairman, Department of Radiology, Albany Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2794
Record Dates: First submitted 2010-09-10; First posted 2010-09-15 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2013-11

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Angioplasty; Vein
MeSH Terms: conditions — Multiple Sclerosis | interventions — Angioplasty; Observation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment of CCSVI with Angioplasty (Experimental): At the time of venography, these patients will have had a significant lesion (blockage) in the internal jugular and/or the azygos vein that will be treated with angioplasty.
  Interventions: Procedure: Angioplasty
- Observation of CCSVI (Sham Comparator): At the time of venography, these patients will have had a significant lesion (blockage) in the internal jugular and/or the azygos vein that will not be treated with angioplasty. These patients will be observed after treatment and compared to those patients who received treatment.
  Interventions: Other: Observation

INTERVENTIONS:
Procedure: Angioplasty — In this procedure, a small catheter (tube) that is approximately the size of a piece of spaghetti is introduced into the vein that is narrowed based on the findings of the venogram. This catheter has a small balloon on it. That balloon is inflated across the narrowing within the vein with the goal of increasing the diameter of that vein and improving flow within that vein.
  Arms: Treatment of CCSVI with Angioplasty
Other: Observation — Patients in this arm will be diagnosed with CCSVI based on venography but will receive no intervention. They will be followed in the same manner as patients treated with angioplasty.
  Arms: Observation of CCSVI

SUMMARY:
The study is being done to determine if venous angioplasty is an effective treatment for chronic cerebrospinal venous insufficiency (CCSVI). In this condition, areas of narrowing or blockages are present in the internal jugular or azygos veins (veins which drain blood from the central nervous system) and these blockages may be associated with symptoms classically attributed to MS. Therefore, angioplasty may help to improve the symptoms associated with CCSVI and multiple sclerosis (MS). In this study, the investigators will evaluate the effectiveness of angioplasty in the treatment of CCSVI by comparing two the outcomes of two groups of patients: one group with CCSVI diagnosed on a venogram and treated with angioplasty and one group with CCSVI diagnosed on a venogram but not treated. The patients enrolled in this study, and the neurologist evaluating patients after the procedure, will not know whether or not they were treated with angioplasty.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are willing to comply with the protocol requirements and can be contacted by telephone
* Patients 18-60 years of age
* Patients with clinically definite multiple sclerosis by Polman criteria
* Patients with a history of MS as defined above with an EDSS between 3-6.
* Patients with a significant stenosis of the internal jugular or azygos vein on the basis of magnetic resonance venography or Doppler ultrasound.

Exclusion Criteria:

* Patients with renal insufficiency based on an estimated GFR <45
* Patients with a known severe allergy to iodine or gadolinium-based contrast agents which cannot be adequately pre-medicated
* Patients with a known allergy to nickel
* Patients who pregnant
* Patients with a contraindication to anticoagulation or anti-platelet medication
* Patients with a contraindication to drugs used for conscious sedation during interventional procedures, including Versed and Fentanyl
* Patients with a history of deep venous thrombosis of the lower extremities
* Patients with occlusion of the right and left common femoral veins
* Patients who have had any changes in their disease modifying drug regimen for MS during the 6 months prior to enrollment in this trial. This would include the addition of any new medications, a change in the dosage of any medications, or the removal of any medications from a patient's drug regimen
* Patients with a life expectancy <18 months
* Patients who are currently enrolled or who plan to enroll in other investigations that conflict with follow-up testing or confounds data in this trial

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2010-08; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Impact of CCSVI treatment on quality of life in patients with MS | 1 Month
  This will be assessed using the Multiple Sclerosis Quality of Life-54 (MSQOL-54), which is a health-related quality of life measure that combines generic and MS-specific items into a single, self-report questionnaire.
Impact of CCSVI treatment on quality of life in patients with MS | 3 Months
  This will be assessed using the Multiple Sclerosis Quality of Life-54 (MSQOL-54), which is a health-related quality of life measure that combines generic and MS-specific items into a single, self-report questionnaire.
Impact of CCSVI treatment on quality of life in patients with MS | 6 Months
  This will be assessed using the Multiple Sclerosis Quality of Life-54 (MSQOL-54), which is a health-related quality of life measure that combines generic and MS-specific items into a single, self-report questionnaire.
Impact of CCSVI treatment on quality of life in patients with MS | 12 Months
  This will be assessed using the Multiple Sclerosis Quality of Life-54 (MSQOL-54), which is a health-related quality of life measure that combines generic and MS-specific items into a single, self-report questionnaire.
Impact of CCSVI treatment on quality of life in patients with MS | 18 Months
  This will be assessed using the Multiple Sclerosis Quality of Life-54 (MSQOL-54), which is a health-related quality of life measure that combines generic and MS-specific items into a single, self-report questionnaire.
Impact of CCSVI treatment on quality of life in patients with MS | 24 Months
  This will be assessed using the Multiple Sclerosis Quality of Life-54 (MSQOL-54), which is a health-related quality of life measure that combines generic and MS-specific items into a single, self-report questionnaire.

SECONDARY OUTCOMES:
Clinical significance of CCSVI in MS patients | 1 month
  This will be assessed clinically using annualized relapse rates, Expanded Disability Status Scale (EDSS) change and change in the timed 25 foot walk.
Superiority of angioplasty to observation for treatment of CCSVI | 1 month
  This will be assessed clinically using annualized relapse rates, EDSS change, and change in the timed 25-foot walk
Incidence of CCSVI in patients with MS | 0 Months
  This will be assessed on the basis of the findings on diagnostic venography of the internal jugular and azygos veins, which is the initial procedure performed in these patients.
Safety of endovascular treatment of CCSVI | 1 month
  This is defined as the number and nature of any procedure-related adverse effects
Target vessel primary and secondary patency | 1 month
  Primary patency is the interval following the initial angioplasty procedure until a reintervention is performed to preserve patency. Secondary patency is defined as the interval following the initial angioplasty procedure until treatment of the vein is abandoned due to an inability to treat the original lesion
Clinical significance of CCSVI in MS patients | 6 months
  This will be assessed clinically using annualized relapse rates, EDSS change and change in the timed 25 foot walk.
Clinical significance of CCSVI in MS patients | 12 months
  This will be assessed clinically using annualized relapse rates, EDSS change and change in the timed 25 foot walk.
Clinical significance of CCSVI in MS patients | 18 months
  This will be assessed clinically using annualized relapse rates, EDSS change and change in the timed 25 foot walk.
Clinical significance of CCSVI in MS patients | 24 months
  This will be assessed clinically using annualized relapse rates, EDSS change and change in the timed 25 foot walk.
Superiority of angioplasty to observation for treatment of CCSVI | 6 Months
  This will be assessed clinically using annualized relapse rates, EDSS change, and change in the timed 25-foot walk
Superiority of angioplasty to observation for treatment of CCSVI | 12 Months
  This will be assessed clinically using annualized relapse rates, EDSS change, and change in the timed 25-foot walk
Superiority of angioplasty to observation for treatment of CCSVI | 18 Months
  This will be assessed clinically using annualized relapse rates, EDSS change, and change in the timed 25-foot walk
Superiority of angioplasty to observation for treatment of CCSVI | 24 Months
  This will be assessed clinically using annualized relapse rates, EDSS change, and change in the timed 25-foot walk
Safety of endovascular treatment of CCSVI | 3 months
  This is defined as the number and nature of any procedure-related adverse effects
Safety of endovascular treatment of CCSVI | 6 months
  This is defined as the number and nature of any procedure-related adverse effects
Safety of endovascular treatment of CCSVI | 12 months
  This is defined as the number and nature of any procedure-related adverse effects
Safety of endovascular treatment of CCSVI | 18 months
  This is defined as the number and nature of any procedure-related adverse effects
Safety of endovascular treatment of CCSVI | 24 months
  This is defined as the number and nature of any procedure-related adverse effects
Target vessel primary and secondary patency | 3 months
  Primary patency is the interval following the initial angioplasty procedure until a reintervention is performed to preserve patency. Secondary patency is defined as the interval following the initial angioplasty procedure until treatment of the vein is abandoned due to an inability to treat the original lesion
Target vessel primary and secondary patency | 6 months
  Primary patency is the interval following the initial angioplasty procedure until a reintervention is performed to preserve patency. Secondary patency is defined as the interval following the initial angioplasty procedure until treatment of the vein is abandoned due to an inability to treat the original lesion
Target vessel primary and secondary patency | 12 months
  Primary patency is the interval following the initial angioplasty procedure until a reintervention is performed to preserve patency. Secondary patency is defined as the interval following the initial angioplasty procedure until treatment of the vein is abandoned due to an inability to treat the original lesion
Target vessel primary and secondary patency | 18 months
  Primary patency is the interval following the initial angioplasty procedure until a reintervention is performed to preserve patency. Secondary patency is defined as the interval following the initial angioplasty procedure until treatment of the vein is abandoned due to an inability to treat the original lesion
Target vessel primary and secondary patency | 24 months
  Primary patency is the interval following the initial angioplasty procedure until a reintervention is performed to preserve patency. Secondary patency is defined as the interval following the initial angioplasty procedure until treatment of the vein is abandoned due to an inability to treat the original lesion

CONTACTS AND LOCATIONS:
Overall Officials: Gary Siskin, MD, Principal Investigator — Albany Medical College
Locations (2):
- United States (2):
  - Albany Medical Center, Albany, New York
  - Image Care Latham, Latham, New York

REFERENCES:
- [Background] Zamboni P, Galeotti R, Menegatti E, Malagoni AM, Gianesini S, Bartolomei I, Mascoli F, Salvi F. A prospective open-label study of endovascular treatment of chronic cerebrospinal venous insufficiency. J Vasc Surg. 2009 Dec;50(6):1348-58.e1-3. doi: 10.1016/j.jvs.2009.07.096. PMID 19958985
- [Background] Zamboni P, Menegatti E, Weinstock-Guttman B, Schirda C, Cox JL, Malagoni AM, Hojanacki D, Kennedy C, Carl E, Dwyer MG, Bergsland N, Galeotti R, Hussein S, Bartolomei I, Salvi F, Zivadinov R. The severity of chronic cerebrospinal venous insufficiency in patients with multiple sclerosis is related to altered cerebrospinal fluid dynamics. Funct Neurol. 2009 Jul-Sep;24(3):133-8. PMID 20018140
- [Background] Bartolomei I, Salvi F, Galeotti R, Salviato E, Alcanterini M, Menegatti E, Mascalchi M, Zamboni P. Hemodynamic patterns of chronic cerebrospinal venous insufficiency in multiple sclerosis. Correlation with symptoms at onset and clinical course. Int Angiol. 2010 Apr;29(2):183-8. PMID 20351674
- [Background] Malagoni AM, Galeotti R, Menegatti E, Manfredini F, Basaglia N, Salvi F, Zamboni P. Is chronic fatigue the symptom of venous insufficiency associated with multiple sclerosis? A longitudinal pilot study. Int Angiol. 2010 Apr;29(2):176-82. PMID 20351673
- [Background] Zamboni P, Galeotti R, Menegatti E, Malagoni AM, Tacconi G, Dall'Ara S, Bartolomei I, Salvi F. Chronic cerebrospinal venous insufficiency in patients with multiple sclerosis. J Neurol Neurosurg Psychiatry. 2009 Apr;80(4):392-9. doi: 10.1136/jnnp.2008.157164. Epub 2008 Dec 5. PMID 19060024